Version 5
EudraCT: 2018-002365-19
Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074
Godkendt LMS: \_\_\_\_\_ Journal nr: 2018061692
Protocol

Testosterone in bariatric patients

27<sup>™</sup> of August 2018

Title

Muscle strength and -mass after bariatric surgery - a possible effect of testosterone replacement therapy?

Randomized, placebo-controlled and double-blinded study

## Research group

Hospital of Southwest Jutland and Odense University Hospital, the Endocrinology units:

Line Velling Magnussen

Hospital of Southwest Jutland, the Endocrinology unit and bariatric team:

Alin Andries, Claus Juhl and Bibi Gram

Odense University Hospital, the Endocrinology unit:

Jeppe Gram, Marianne Andersen, Dorte Glintborg and René Støving

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074
Godkendt LMS: \_\_\_\_\_ Journal nr: 2018061692

# TABLE OF CONTENTS

| 1. GENERAL INFORMATION | 3 |
|-------------------------------------------|----|
| 2. INTRODUCTION | 5 |
| 3. TRIAL PLAN AND DESIGN | 7 |
| 4. STUDY POPULATION | 9 |
| 5. TREATMENT OF PATIENTS | 10 |
| 6. EVALUATION OF EFFECT | 13 |
| 7. SAFETY | 16 |
| 8. STATISTICS | 17 |
| 9. SOURCE DATA | 18 |
| 10. QUALITY CONTROL AND QUALITY ASSURANCE | 18 |
| 11. ETHICAL QUESTIONS. | 18 |
| 12. HANDLING AND ARCHIVING DATA | 19 |
| 13. BIO BANK | 20 |
| 14. FINANCING AND INSURANCE. | 20 |
| 15. GUIDELINES FOR PUBLICATION. | 20 |
| 16. SUMMARY AND APPENDICES | 20 |
| 17. LITERATURE REFERENCES. | 21 |
| APPENDIX | 24 |

EudraCT: 2018-002365-19

27<sup>™</sup> of August 2018

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: Journal nr: 2018061692

#### 1. General information

Sponsor, primary, practical and coordinating investigator:

Line Velling Magnussen, MD, PhD

Phone: 29787835

E-mail: line.velling.magnussen@rsyd.dk

### Investigators:

Hospital of Southwest Jutland (SVS) and Odense University Hospital (OUH), the Endocrinology units:

Line Velling Magnussen

Hospital of Southwest Jutland, the Endocrinology unit and bariatric team

Haraldsgade 7F, 6700 Esbjerg:

Alin Andries, Claus Juhl and Bibi Gram

Odense University Hospital, the Endocrinology unit

Kløvervænget 6, 5000 Odense:

Jeppe Gram, Marianne Andersen, Dorte Glintborg and René Støving

The trial will be monitored in accordance with GCP, and the local GCP unit will help establish the extent of the monitoring to ensure that the trial comply with GCP and applicable law. The trial will be conducted according to this protocol. The study protocol will be submitted to The Danish Medicines Agency and the Regional Ethics Committee, notified to the Danish Data Protection Agency and registered at ClinicalTrials.gov. The investigations are conducted as part of a post.doc position at the University of Southern Denmark.

### Collaborators:

KBA at SVS and OUH (biochemistry)

Institute of Regional Health Research/Centre of Southwest Jutland (muscle strength and VO2max)

Physical Therapy section (exercise counseling)

The GCP-section at Odense University Hospital

OPEN (randomization and eCRF)

Pharmacy at OUH (handling of study medicine)

| Version 5 EudraCT: 2018-002365-19 Godkendt VEK: Projekt ID: S-20180074 Godkendt LMS: Journal nr: 2018061692 | 27 <sup>™</sup> of August 2018 |
|---|---|
| Time schedule: | |
| Estimated August 2018 – January 2021 | |
| Sponsor, primary, practical and coordinating investigator: | |
| Line Velling Magnussen, MD, PhD | |
| Hospital of Southwest Jutland and Odense University Hospital, the Endocrinol- | ogy units. |
| Phone: 29 78 78 35. | |
| E-mail: Line.velling.magnussen@rsyd.dk | |

Signature

Date

EudraCT: 2018-002365-19

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: Journal nr: 2018061692

#### 2. Introduction

Obesity, poor physical fitness and low muscular strength are associated with all-cause mortality [1-5]. Loss of bodyweight is commonly achieved by diet with or without exercise intervention. However, both diet and diet+exercise programs are often followed by weight regain and it is generally difficult to achieve long-term weight loss [6].

There are many challenges associated with the counselling of obese and sedentary individuals in order to increase their physical activity (PA), and there may be a need for a tight schematic counselling to achieve positive results [7]. Additionally, promoting PA among patients that have undergone bariatric surgery has also shown to be challenging [8, 9] even though PA may be of a great importance regarding several postoperative outcomes [9-12]. Lifestyle changes following bariatric surgery may be important for the overall effect of the BS in the long term. Therefore, it is vital to find an appropriate and well-suited setting to improve PA among these patients. When structuring PA counselling, the five A's (Assess, Advise, Agree, Assist, Arrange) might be a helpful tool and it is considered important to engage the patients in PA counselling both before and after the surgery [9, 13].

Loss of bodyweight reduces morbidity and mortality [14]. Bariatric surgery is the most effective method to treat severe obesity and type 2 diabetes mellitus achieving high remission rates [15]. However, weight loss also decreases skeletal muscle mass [16, 17] which might counterbalance the positive effects of a bariatric surgery since low lean body mass is linked to increased mortality under various circumstances (i.e., heart disease, cancer, burn injuries) [18]. Furthermore, a substantial loss of bone mass is seen after bariatric surgery [19, 20] despite weight stability in the second-year post-operative [19], which could have important clinical implications for long-term skeletal health with increased fracture risk [19, 21]. On the other hand, the loss of muscle and bone mass could merely be a natural adaptation to a lower weight after bariatric surgery. Studies trying to establish whether the loss of muscle mass is disproportionately in patients following bariatric surgery compared to BMI-matched controls are conflicting, showing lower muscle mass in both sexes after surgery compared with their respective matched controls assessed by magnetic resonance imaging in one study [22] whereas another study has shown comparable fat-free mass 24 months post-operative assessed by bioelectric impedance [23]. Currently, there are no effective approaches to prevent the immense loss of muscle and bone mass following bariatric surgery [18] although several approaches can be considered, e.g. exercise and dietary intervention [24].

EudraCT: 2018-002365-19 27<sup>TH</sup> of August 2018

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: \_\_\_\_\_ Journal nr: 2018061692

Low testosterone levels have been associated with sarcopenia, insulin resistance, increased body fat, reduced quality of life and loss of libido and sexual function. Testosterone therapy increases lean body mass (i.e. muscle mass), improves bone density and decreases fat mass [25]. As up to 78.8% of patients undergoing bariatric surgery suffer from low testosterone levels [26-28], testosterone therapy prior to and after bariatric surgery may prevent or reduce the considerable loss of muscle mass during the weight loss period [29]. So far, no studies have evaluated the effect of testosterone therapy combined with exercise and diet counselling on body composition and quality of life in men undergoing bariatric surgery.

# Testosterone therapy and cardiovascular risk

Studies on cardiovascular risk during testosterone therapy are conflicting. A study in old men with limitations in mobility showed significantly more cardiovascular events during testosterone therapy compared to placebo and the study was ended prematurely [30]. Low HDL levels are linked to an increased morbidity and mortality of cardiovascular disease. A significant small decrease in HDL cholesterol levels in men treated with testosterone was reported in a meta-analysis [31] and a systematic review [32]. However, a large observational study on pooled data in obese, hypogonadal diabetic men during six years of testosterone therapy reported a favorable change in lipid profile along with reduced pulse pressure and reduced arterial stiffness, which are independent risk factors for cardiovascular disease [33]. Another approach in clarifying the effect of testosterone therapy on cardiovascular disease risk is the evaluation of biomarkers for cardiovascular disease during therapy, i.e. soluble Klotho, a protein, which may function as a hormone [34]. Higher levels of soluble Klotho are independently associated with a lower likelihood of having cardiovascular disease [35]. To date, no reports on Klotho have been published in obese patients undergoing bariatric surgery during testosterone therapy.

Few studies have addressed the influence of testosterone therapy on the haemostatic system. Thrombin generation (TG) measures are risk markers of cardiovascular disease and address the composite of multiple factors that influence blood coagulation [36]. One intervention study showed that i.m. testosterone treatment for one year in elderly men with low testosterone levels had no impact on thrombin generation measured at one year [37]. A significant number of patients sustaining venous thrombotic events after initiation of testosterone therapy often had inherited cardiovascular risk factors such as Factor V Leiden [38], and thrombotic events were primarily

EudraCT: 2018-002365-19

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074

Godkendt LMS: Journal nr: 2018061692

observed within the first months of testosterone treatment, suggesting that testosterone therapy triggers cardiovascular events in thrombosis prone individuals. Thus, studies on both the short term and the long term impact of testosterone treatment on the haemostatic system are warranted [38, 39].

## Pseudo-Cushing's syndrome

Central obesity results in a cluster of metabolic abnormalities contributing to premature death, socalled Pseudo-Cushing's syndrome [40]. Glucocorticoids regulate adipose-tissue differentiation, function and distribution, and in excess, cause central obesity. To our knowledge, no studies have reported results on levels of cortisol and testosterone before and after bariatric surgery.

# 3. Trial plan and design

#### General aim

To investigate the effect and clinical relevance of testosterone therapy combined with exercise and diet counselling in hypogonadal men undergoing bariatric surgery.

### **Objectives**

To evaluate the effect of testosterone therapy combined with exercise and diet counselling on muscle strength, body composition, hormones, components of the metabolic syndrome, inflammation, sexual function, and quality of life after weight loss in obese, hypogonadal men undergoing bariatric surgery.

### **Perspective**

The study will investigate whether testosterone therapy can stabilize muscle function, prevent the substantial decrease in muscle mass (lean body mass), and improve components of the metabolic syndrome, inflammation and quality of life in patients after bariatric surgery.

### Study design

A two centre, randomized, double-blind, placebo-controlled study on testosterone therapy combined with lifestyle intervention, in men eligible for bariatric surgery with low testosterone levels. Routine

EudraCT: 2018-002365-19 27<sup>TH</sup> of August 2018

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: \_\_\_\_\_ Journal nr: 2018061692

bariatric procedure will be conducted between 3 and 6 months after inclusion. The end of the study is 52 weeks postoperatively.

## Study endpoints

## Primary outcome:

- Maximal isometric muscle strength (N) in shoulder muscles (shoulder elevation.

## Secondary outcomes:

- Regional body composition (DXA scan, BMI, Waist/hip-ratio)
- Physical strength: maximal isometric muscle strength in lower extremities (hip extension, hip abduction), muscle strength in upper-extremities (shoulder abduction, shoulder adduction)
- Physical function: performance-based measures of physical function (stair climb test) and maximal oxygen uptake (VO<sub>2</sub>max).
- Glucose metabolism (HOMA-R, HbA1c, Fasting-P-Blood glucose)
- Coagulation/fibrinolysis status (thrombin generation measures)
- Adipokines and inflammation markers (leptin, adiponectin, hsCRP, IL-6, suPAR, lipid profile (HDL, LDL, triglycerides))
- Hormones and binding proteins (testosterone, SHBG, LH, FSH, prolactin, CBG, growth hormone-axis (IGF-I and IGF-II, IGFBPs, bioactive IGF-I), cortisol, aldosterone, Cortisol and cortisol metabolites)
- Vascular markers (soluble Klotho, fibulin-1)
- Bone markers and calcitropic hormones (osteocalcin, PINP, 1CTP, CTX, PTH, 25OH-vitaminD, 1.25(OH)2-Vitamin-D)
- Quality of life and sexual function (International Index of Erectile Function (IIEF-5), Major Depression Inventory (MDI), World Health Organization Well Being Index (WHO-5), Physical function component of Vitality scale of Short Form 36 (SF36)

EudraCT: 2018-002365-19

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: Journal nr: 2018061692

#### Method

A randomized, double-blind, placebo-controlled intervention study in men eligible for bariatric surgery and low testosterone levels (total testosterone < 12.0 nmol/l [41]). Routine bariatric procedure will be conducted between 3 and 6 months after inclusion.

### 4. Study population

#### Recruitment

Patients will be recruited among bariatric patients at Hospital of Southwest Jutland and at Odense University Hospital. As part of a review of existing clinical practice in the Region of Southern Denmark, patients who are entitled to bariatric surgery are currently subject to an audit with the establishment of a quality and research database. As part of the audit, patients have had their testosterone levels in the blood measured. MD Line Velling Magnussen (LVM) may obtain these results from the journal, if there is a signed consent statement during the audit, where the patients also have agreed to be contacted for future projects, where their participation will be relevant. MD LVM may phone those patients with low testosterone levels and send the written information regarding the trial along with the booklets "Før du beslutter dig" and "Forsøgspersoners rettigheder i et sundhedsvidenskabeligt forskningsprojekt", if agreed by the patients. Patients are informed that they are entitled to bring a bystander for the oral information. Those who may wish to participate, are contacted on the first day of the participation of the patient school at the Southwest Hospital of Jutland, Esbjerg (as part of the standard treatment procedure prior to bariatric surgery), where a MD from the research team, all of whom have experience within the field of bariatri and GCP experience, will provide oral information regarding the trial. The information is giving in a suitable room, ensuring that the conversation can take place without interference. After the oral information, the patient has minimum 24 hours to think about participation. Upon acceptance, time is given for visits, screening blood samples and obtaining written informed consent. Inclusion will be in the beginning of the mandatory 8% weight loss period lasting 3-6 months.

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: Journal nr: 2018061692

#### Overview:



### Randomization

After the baseline assessment, the patients will be randomly assigned to either testosterone or placebo. The randomization sequence will be created using OPEN Randomise, stratifying patients with a 1:1 allocation using random block sizes of 2, 4 and 6. The allocation sequence will be concealed from the researcher enrolling and OPEN Randomise will send an e-mail to an email address each time a randomization is performed.

#### Inclusion criteria

- Eligible for bariatric surgery according to the Danish national criteria (i.e. aged 18–60 years, BMI >35 kg/m2 with specific secondary disease or BMI >40 kg/m2 with significant health issues assessed by the multidisciplinary bariatric team) [42]
- Caucasian men
- Total testosterone < 12.0 nmol/l
- No contraindications for testosterone treatment

#### **Exclusion criteria**

- Previously diagnosed with prostate, mammae or liver cancer. Any other cancer within the last 5 years.
- Hypersensitivity to the active substance or to any of the excipients in Nebido<sup>®</sup>
- Symptomatic heart disease NYHA >2
- Recently thromboembolic disease <3 months
- PSA >4.0 ug/l or PSA>3.0 ug/l and lower urinary tract symptoms
- Disability that severely affect the ability to perform exercise training
- EVF > 52%

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074
Godkendt LMS: \_\_\_\_ Journal nr: 2018061692

The following treatments are not allowed in the study

- 5-α-reductase inhibitors

- Prednisolone >5mg/day

## 5. Treatment of patients

## **Treatment regimen**

- Inj. Testosterone undecanoat (Nebido®), 1000 mg im or placebo preoperative (baseline, weeks 6, 18 and 30 depending on time to surgery) and postoperative (weeks 4, 16, 28, 40) (Table 1).
- Administration: deep and slow (over two minutes) intragluteal injection
- Due to the risk of anaphylaxis, patients are observed at least 30 minutes on the test site after the first two injections

## Non-pharmacological intervention

- Routine bariatric procedure (Roux en Y gastric bypass or sleeve gastrectomy). Surgery will be conducted between 3 and 6 months after inclusion.
- Lifestyle intervention program: Routine instructions on diet and dietary precautions after surgery [43] and individual exercise counseling three times after surgery.

## Contraindications Testosteron undecanoate (ATC-code G03BA03)

- previously diagnosed with prostate, mammae or liver cancer. Any other cancer within the last 5 years.
- hypersensitivity to the active substance or to any of the excipients

### Caution in

- cardiac insufficiency, especially known ischemic heart disease and hypertension
- hepatic or renal insufficiency
- clotting disorders / anti-coagulant treatment
- known epilepsy and migraine
- pre-existing sleep apnoea

EudraCT: 2018-002365-19

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074
Godkendt LMS: \_\_\_\_ Journal nr: 2018061692

Adverse reactions (see Appendix).

Study medicine is administered at the departments of endocrinology at SVS or OUH. Study medicine is handled according to annex 13.

Patients are treated with Testosterone Undecanoate 1000 mg/4 ml, intramuscular (i.m.) or placebo. Study medicine and placebo have been produced by Bayer Health Care. Packing, blinding, labeling and randomization of study medicine are done by the pharmacy of Odense University Hospital according to annex 13: Name of sponsor, route of administration, batch number, trial reference code, user manual for study medicine, storage of study medicine expiration date (a copy of the label is placed in the trial master file).

The medicine (active and placebo) is delivered to the pharmacy from Bayer with no labels. Identical labels will be put on the ampules, with the exception of the randomization number.

Study medicine can be used only in clinical trials.

Sponsor is responsible for the destruction of surplus medicine.

#### **Medicine records**

All medicine is accounted for in total and for every patient. The records are kept in the trial master file. The randomization code is kept according to law. The procedure for code breakage: In case of a medical emergency an investigator is allowed to break code and inform whether testosterone or placebo is administered. Other members of the study group will remain blinded. The patient will be excluded from the study if the code is broken. Testosterone treatment is a registered treatment. It is not of clinical significance for further acute treatment to know within 24 hours if a patient is in active treatment or not. All the investigators who are medical doctors are affiliated with one the departments of endocrinology at SVS or OUH. At least one of these investigators has their cell phone open 24 hours a day, also during vacations.

### Discontinuation of study treatment

Treatments stop:

- Confirmed increase in serum PSA > 3 ug/l and clinical symptoms and at least 20% increase since baseline is followed by referral to urological evaluation
- Suspicion of prostate cancer

EudraCT: 2018-002365-19 27<sup>TH</sup> of August 2018

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: \_\_\_\_\_ Journal nr: 2018061692

- Hematocrit (EVF) > 0.52 and at least 20% increase since baseline
- Serum ALAT >3 times upper normal limit and at least 20% increase since baseline
- Patients can leave the study prior to end of study, due to safety issues (increased safety parameters), fulfillment of exclusion criterion, at own request or due to lack of compliance including failure to achieve 8% weight loss prior to operation.

#### **Pharmacokinetics**

Nebido® slowly releases testosterone after intramuscular injection with no first-pass effect. Testosterone is metabolized in the liver (CYP3A4) to active metabolites estradiol and dihydrotestosterone. An increase in serum levels of testosterone above basal values may be seen one day after administration, and has an average half-life time of 50-130 days. Steady-state conditions are expected to be achieved between the 3rd and the 5th administration with constant dosing interval of 10 weeks during the following administrations. The median intra- and interindividual variability (coefficient of variation, %) of Cmin values was 22 % (range: 9-28%) and 34% (range: 25-48%), respectively.

EudraCT: 2018-002365-19

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: Journal nr: 2018061692

### 6. Evaluation of effect

Assessments according to visits:

| Table 1 | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Pre-operative | | | Per/Post-operative | | | | | | |
| | Baseline | W | W | W | W | W | W | W | W | W |
| | | 6 | 18 | 30 | 0 | 4 | 16 | 28 | 40 | 52 |
| Testosterone injection* | X | X | X | X | | X** | X | X | X | |
| Safety | X | X | X | | X | | X | X | | X |
| Exercise and diet counseling | X | | | | X | | | X | | X |
| Muscle strength and VO <sub>2</sub> max test | X | | | | X | | | X | | X |
| Physical examination | X | | | | X | | | X | | X |
| Blood samples | X | | | | X | | | X | | X |
| Urine samples | X | | | | X | | | | | X |
| Body composition (DEXA scan) | X | | | | X | | | X | | X |
| Questionnaires | X | | | | X | | | X | | X |
| Dexamethasone suppression test | X | | | | X | | | | | X |

W=weeks, W0= from one to seven days before operation.

## **Blood samples**

- 1) Hormones and binding proteins: Total testosterone, SHBG, LH, FSH, prolactin, CBG, growth hormone-axis (IGF-I and IGF-II, IGFBPs, bioactive IGF-I), cortisol, ACTH
- 2) Adipokines and inflammation markers (leptin, adiponectin, hsCRP, IL-6, suPAR, YKL40, GDF15, sCD36, FGF23, phosphate, total-calcium, lipids)

<sup>\*</sup> Number of injections depends on time to achieve the mandatory 8% preoperative weight loss. The testosterone injection needs to be applied in the preoperative period at Weeks 6 and hereafter every 12 weeks, correspondingly Weeks 18 and Weeks 30 if necessary.

<sup>\*\*</sup> The first time for injection in the postoperative period will be 12 weeks after the last injection during the preoperative period. Injection within 4 weeks before planned surgery is postponed to week 4 +/- 2 weeks postoperatively.

EudraCT: 2018-002365-19 27<sup>TH</sup> of August 2018

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074
Godkendt LMS: \_\_\_\_ Journal nr: 2018061692

- 3) Vascular markers (aldosterone, fibulin-1, soluble Klotho)
- 4) Bone markers and calcitropic hormones (osteocalcin, PINP, 1CTP, CTX, PTH, 25OH-vitaminD)
- 5) Glucose metabolism: s-insulin, HbA1c, Fasting-P-Blood glucose
- 6) Safety parameters (hemoglobin, hematocrit, PSA, ALAT)
- 7) Coagulation/fibrinolysis status (thrombin generation measures)

# **Urine samples**

Diurnal U-Cortisol and cortisol metabolites

## **Body composition**

Whole body composition, lumbar and hip bone mineral density and will be assessed using Dual x-ray absorptiometry (DEXA) on Hologic Discovery devices (Waltham, MA, US). DXA scans will be performed at the Department of Endocrinology, SVS.

## Questionnaires

The participants will be asked to fill in standardized and validated questionnaires regarding quality of life and sexuality:

- Short Form 36 (SF-36) from Qualimetrics (qualimetrics.com)
- IIEF5 –International Index of Erectile Function, copyright of Pfizer Danmark, Lautrupvang 8, 2750 Ballerup
- Major Depression Inventory (MDI)
- World Health Organization Well Being Index (WHO-5)

# Dexamethasone suppression test

The test is used in diagnosing Cushing's syndrome by measuring how cortisol levels change in response to 1 mg dexamethasone overnight.

EudraCT: 2018-002365-19

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: Journal nr: 2018061692

#### Physical examination

- 1) Body weight: will be measured on calibrates scales with patients only wearing their underwear (no shoes)
- 2) Height: will be measured without shoes
- 3) BMI will be calculated by the formula weight/height<sup>2</sup> (kg/m<sup>2</sup>)
- 4) Waist: will be measured in the middle of the distance between the 12th rib and antero-superior iliac spine, while keeping the measuring tape parallel with the floor
- 5) Hip: will be measured across the widest part of the hips while keeping the tape parallel to the floor
- 5) Waist/hip ratio will be computed
- 6) Blood pressure measures thrice while sitting (the participants are to be seated at least 5 minutes prior to the measurements). The mean of the last two measurements is registered
- 7) Testicular volume will be assessed by using Prader orchid meter
- 8) Changes in primary and secondary sex characteristics (breast size / gynecomastia and pubic hair) will be assessed by using the Tanner scale

#### Muscle strength testing

- 1) Muscle strength: Maximal isometric muscle strength will be measured with a Bofors MODEL dynamometer (Bofors Elektronik, Karlskoga, Sweden). Three maximal voluntary contractions (MVC) with 30 seconds of recovery between attempts will be conducted, and the highest value will be recorded. Maximal force and the corresponding moment arm will be registered [44].
- 2) VO2 max and functional capacity: Maximal oxygen uptake will be estimated from the relation between sub-maximal workload and stable heart rate obtained in Astrand one-point sub-max test [45]. The bike test will be conducted by using Monark 939E electronic ergometer work test bike (939E) which is digitally controlled and has embedded protocol and calculation of max VO2 (Astrand formula). The pedaling frequency will be adjusted at 60 rounds per minute and the initial workload is 450 kilopond meter/minute (corresponding to ~ 75 watt).
- 3) Functional capacity will be estimated using stair-climb test. The outcome is the number of times the subjects are able to reach the stairs up and down for a period of one minute.

EudraCT: 2018-002365-19

2018-002365-19

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074
Godkendt LMS: Journal nr: 2018061692

7. Safety evaluation

Monitoring:

- Physical examination (baseline, per/postoperative weeks 0, 28 and 52) (Table 1)

- Biochemical examinations: 1. testosterone levels (baseline) 2. PSA, EVF, ALAT (baseline,

preoperative weeks 6 and 18, postoperative weeks 0, 16, 28 and 52)

- Clinical relevant abnormal measurements are repeated

Safety parameters:

- Measurements of hematocrit: testosterone therapy increases the hematocrit level and high

levels of hematocrit leads to higher risks of venous thrombosis (Danish Urological Society

(DUS) 2013).

- In order to take into account the Danish Urology Cancer Group (DUCG) 2013 report on

prostate cancer, and the Danish Urological Society report on androgen substitution (2013)

the exclusion criterion for PSA in the study is based on the above level.

Registration and reporting of adverse events:

An adverse event: Any untoward medical occurrence in a patient or clinical trial subject

administered a medicinal product and which does not necessarily have a causal relationship with

this treatment.

A serious adverse event: Any untoward medical occurrence or effect that at any dose results in

death is life threatening, requires hospitalization or prolongation of existing hospitalization, results

in persistent or significant disability or incapacity, or is a congenital anomaly or birth defect. All

serious adverse events are reported from investigator to sponsor within 24 hours of becoming

aware.

Adverse events are reported to Danish health and medicines authority and regional ethics committee

according to current guidelines. Other investigators are informed.

The sponsor ensures that all relevant information about suspected unexpected serious adverse

reactions (SUSARs) that are fatal or life threatening is recorded and reported as soon as possible to

the competent authorities and to the Ethics Committee no later than seven days after knowledge by

the sponsor of such a case. Relevant follow-up information is subsequently communicated within

an additional eight days.

17

EudraCT: 2018-002365-19

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074
Godkendt LMS: Journal nr: 2018061692

27<sup>™</sup> of August 2018

All other suspected serious unexpected adverse reactions will be reported to the Danish health and medicines authority (DKMA) and to the Ethics Committee concerned as soon as possible but within a maximum of 15 days of first knowledge by the sponsor. The sponsor is obliged to inform all investigators.

A definition of a suspected unexpected serious adverse reaction (SAR) is as follows: An adverse reaction, the nature or severity of which is not consistent with the applicable product information as not being according to the summary of product characteristics of Nebido®. The reference document used is the specified product summary for Nebido® (section 4.8 of the summary), when assessing whether a SAR is unexpected/expected, thus possibly becoming a SUSAR.

SUSARs are reported electronically (e-blanket) to DKMA.

All adverse events are registered. Sponsor is obliged to report a list of serious adverse events to DKMA and the regional ethics committee annually.

Sponsor will forward serious adverse events and suspected unexpected serious adverse reaction to Bayer within 24 hours of becoming aware.

Treatment of complications and follow-up:

- Patients will be referred to the relevant specialist department for further control and possible treatment.

Criteria for end of study:

- The study will end after 52 weeks of testosterone therapy postoperatively. The patients will be offered a visit in the clinic six months after end of study.
- Patients can leave the study prior to this due to safety issues (increased safety parameters), fulfillment of exclusion criterion, at own request or due to lack of compliance including failure to achieve 8% weight loss prior to operation.

### 8. Statistics

Sample size: The power and sample size calculation is based on the primary outcome maximal voluntary isometric contraction in shoulder muscles (shoulder elevation) after the intervention. To detect a minimal relevant difference between (MIREDIF) of 14% [46] the groups with a two-sided significance level of 0.05 assuming a SD of 34 N [46], and to obtain a power 80%, it is required to

EudraCT: 2018-002365-19

2010-002505-19

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: \_\_\_\_\_ Journal nr: 2018061692

enroll 18 patients in the ITT-population. We will include 25 participants in each group to account for drop outs.

Statistical analyses: All data being collected, primary and secondary outcomes will be analyzed according to the ITT principle. Missing data were handled by multiple imputations, assuming missing values were randomly distributed. Baseline demographic and clinical characteristics will be reported descriptively for all patients in the full analysis set. For assessments of change from baseline, analyses of covariance (ANCOVA) will be applied, with treatment assignment serving as the main factor and the baseline value as covariate. Unless stated otherwise, results will be expressed as the difference between the group means with 95% confidence interval. P values will be reported if appropriate. Significance level: 5%. Additionally to the ITT analyses per protocol analyses will be conducted.

### 9. Source data

Source data includes patient journals and laboratory/scan reports using eCRF in REDCap through OPEN. Direct access to source data is allowed in monitoring of the study, audit and inspection from ethics committee, Danish health and medicines authority, the Danish data protection agency and other relevant health authorities. This is accepted by participants in a written authorization.

## 10. Quality control and quality assurance

Quality control and securing of quality is done according to §§ 3 and 4 in the GCP–guidelines, annex 3 and GCP guidelines section 1.46 and 1.47.

### 11. Ethical questions

An increasing number of patients become obese. Bariatric surgery is an effective method in the treatment of severe obesity and T2D achieving high remission rates. However, weight loss also decreases skeletal muscle mass. Obesity together with poor physical fitness and low muscular strength is associated to all-cause mortality. As many patients undergoing bariatric surgery suffer from low testosterone levels, testosterone therapy may prevent the immense loss of muscle mass together with physical and diet counselling in these patients. So far, no other treatment has prevented this loss of muscle mass. Hence a study like this is needed to investigate if testosterone therapy in these patients will be beneficial.

EudraCT: 2018-002365-19

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: \_\_\_\_\_ Journal nr: 2018061692

Nebido® is registered in Denmark. Injection with testosterone or placebo can be uncomfortable for some. The drug is administered in the gluteal muscle and local swelling and redness of the skin can be observed. This is temporary and safe. The study is in accordance with the Helsinki II declaration and is reported to the regional ethics committee and the Danish health and medicines authority. Individuals found eligible to bariatric surgery and who accept to undergo the operation will be included in the study at the beginning of the mandatory 8% preoperative 6 month's weight loss period. Individuals will be recruited among patients referred to bariatric surgery at Hospital of Southwest Jutland and at Odense University Hospital. Patients will be asked at their first attendance at the clinic if they would like to consider participation in the study and if so they will receive written information regarding the study and they will be contacted by MD Line Velling Magnussen. It will be emphasized that participation is voluntary and that the consent can be withdrawn at any time and that this will not have any relevance further treatment. The written information concerning the trial will follow guidelines regarding information and consent requirements. All patients will be provided written information material (see appendix). For oral information, this will include an explanation of the written information and a further description of the study. Information relating to patients is protected by the law on the processing of personal data and the law on patients' legal status.

In this trial, half of the patients are treated with Nebido®, which is an approved and marketed testosterone product. The other half will receive injection with placebo. Placebo is necessary during this double-blinded study for methodological reasons. It could affect the results of the trial, if the patients or healthcare staff know in advance whether active treatment is given or not. As always, in clinical trials, unknown effects or complications might occur. Patients cannot be guaranteed effect of treatment, but it is highly probable that: The patients randomized to Nebido® experience an improvement in their muscle mass and muscle strength, as well as improved quality of life and reduced symptoms associated with low testosterone levels. The patients randomized to placebo will receive counseling in relation to exercise before and after bariatric surgery compared to standard procedure. As standard treatment is used as comparative treatment, no one is treated differently or worse compared to the normal treatment procedure, including standard follow-up by physician, dietitians and nurses in the clinic. The knowledge gained through the experiment will contribute with significant scientific information of importance to the future treatment of men undergoing bariatric surgery. Thus, it is the opinion of the investigators that the trial is relevant and ethical.

EudraCT: 2018-002365-19

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: \_\_\_\_\_ Journal nr: 2018061692

The DXA scans in the study program give rise to a radiation dose of 1 mSV, which corresponds to 1/7 of the background radiation per year in Denmark. Exposure for 1 mSv increases the risk of dying of cancer by 0.005%. The background risk of dying of cancer in Denmark is 25%. Participation in the project will mean exposure to ionizing radiation for patients, which will give rise to a risk increase from 25% to 25.00125%. This does not affect current or future health. The patients will be offered a visit in the clinic six months after end of study including a physical examination and control of androgen status.

# 12. Handling and archiving data

Data is handled and filed according to EMEA guidelines for Good Clinical Practice section 5.5.

Data is collected and analyzed electronically (OPEN) and no unauthorized access to data is allowed.

Original data is filed according to one participant number.

The study is reported to the Danish Data Protection Agency (joint report from the Region of Southern Denmark) and will be handled according to the regulations of the Act on Processing of Personal Data. Data will be stored for 10 years.

This is a privately initiated trial and hence sponsor is responsible for data. Information on concomitant medication and patient history from the medical journal will be given to the investigator as part of the inclusion procedure to secure that the exclusion criteria are met and later on for the evaluation of the effect of testosterone therapy in patients undergoing bariatric surgery. In the latter case referring to data observed during the study: physical examination (weight, height, hip goal, waist circumference, breast development, blood pressure), blood tests and urine tests.

### 13. Bio bank

A research bio bank will be established for blood (approximately 200 ml) and urine (approximately 300 ml) per participant. The purpose is to analyze blood and urine according to section 6 as part of this trial. Some of the analyses will be conducted during the trial due to evaluation of "safety", lack of resistance to freezing or as part of everyday analyses, whereas other analyses will be performed after end of trial due to economic and/or methodological reasons. If the research group wishes to carry out other analyzes than those approved in the current project material, the Regional Ethics Committee must be requested for permission. After the study is finished, the remaining material will be fully anonymized and kept for 10 years and then destroyed.

EudraCT: 2018-002365-19

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: \_\_\_\_\_ Journal nr: 2018061692

## 27<sup>TH</sup> of August 2018

# 14. Financing and insurance

Investigator initiated research project. Funding is obtained from Hospital of Southwest Jutland, Odense University Hospital and Region of Southern Denmark. The investigators and the departments of endocrinology have no financial gain regarding the study and no conflict of interest that could be perceived as prejudicing the impartiality of this study. The patients will not receive payment. The placebo and Nebido have been donated by Bayer. There will be applied for additional research grants.

The study is conducted under the insurance of the department of endocrinology, SVS.

The grant from the Region of Southern Denmark has been placed on a project account by Deputy Head in "økonomi og planlægning" Morten Lyhne Jørgensen at the Hospital of Southwest Jutland. Sted no. 101 123 190 123. Account 138 61 633 04.

### **Budget**

| | Støtte opnået fra | _ | Opnået støtte fra anden | | Total budget i perioden |
|---|---|---|---|---|---|
| | bevilling fra Region | | steds til brug i perioden | andet steds | |
| | Syddanmarks | ansøgte periode | | | |
| | Forskningspuljer | | | | |
| LØN | | | | | |
| Videnskabeligt personale | | | | | |
| Postdoc (20%) | | | 402.000 | | 402.00 |
| Videnskabelige medarbejdere SVS | | 402.000 | | | 402.00 |
| Videnskabelige medarbejdere OUH | | 201.000 | | | 201.00 |
| Teknisk administrativt personale | | | | | |
| Forskningssygeplejersker | 200.000 | | | 70.000 | 270.00 |
| DRIFT | | | | | |
| Dexa-skanning, blodprøver, urinprøver | 800.000 | | | 250.000 | 1.050.00 |
| UDSTYR -APPARATUR | | | | | |
| Andet | | | | | |
| Medicin | | | 375.000 | | 375.00 |
| Overhead (3,1% ) af totale omkostninger | | | | | |
| TOTAL | 1.000.000 | <b>603.000</b> | 777.000 | 320.000 | |
| Țotal budget | | | | | 2.700.00 |
| Forklarende tekst til budget og de | enkelte hudget | tnoster: | | | Ĭ |
| | • | • | mmatian markare 1 | /accular markors D | |
| Blodprøver: Hormones and bindin | | | • | | |
| markers and calcitropic hormones | • | olism, Safety pa | rameters , Coagulat | ion/fibrinolysis stat | us. Se |
| venligst ansøgning for nærmere s | pecifikation. | | | | |
| Urinprøver: diurnal U-Cortisol and | l cortisol metabo | olites | | | |
| Medicin: Dexametason, Nebido/p | lacebo | | | | 0 |

### 15. Guidelines for publication

EudraCT: 2018-002365-19 27<sup>TH</sup> of August 2018

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: \_\_\_\_\_ Journal nr: 2018061692

The study is registered at clinicaltrials.gov and publication is according to the Vancouver regulation.

The study group is obliged to publish positive, inconclusive as well as negative results. Sponsor will inform the Danish medicines agency no later than 90 days after study end and 1 year after study end report study outcomes to the Danish medicines agency (lov om lægemidler § 89, stk. 2, nr. 4). In summarized form: number of treated patients, used doses, results and adverse events. The Danish medicines agency can ask for the full study report.

# 16. Summary and appendices.

#### Resume

Bariatric surgery is an effective method in the treatment of severe obesity and type 2 diabetes mellitus achieving high remission rates. However, weight loss also causes loss of skeletal muscle and bone mass which at least partly could be prevented by exercise and dietary intervention although the counselling of obese and sedentary individuals in order to increase their physical activity presents a challenge. As up to 78.8% of men undergoing bariatric surgery have low levels of testosterone, testosterone therapy could be considered an attractive alternative or supplement to prevent the immense loss of muscle mass during weight loss. Furthermore, low testosterone levels are associated with sarcopenia, insulin resistance, increased body fat, reduced quality of life, loss of libido and reduced sexual function. The study is a long-term randomized, placebo-controlled trial investigating the effects of testosterone therapy combined with exercise and diet counselling on body composition, components of the metabolic syndrome, hormones, inflammation, sexual function and quality of life before and after weight loss in obese, hypogonadal men undergoing bariatric surgery.

#### 17. Literature references

- 1. Ruiz JR, Sui X, Lobelo F, Morrow JR, Jr., Jackson AW, Sjostrom M, Blair SN: **Association between muscular strength and mortality in men: prospective cohort study**. *BMJ (Clinical research ed)* 2008, **337**:a439.
- 2. Laukkanen JA, Rauramaa R, Salonen JT, Kurl S: **The predictive value of cardiorespiratory fitness combined with coronary risk evaluation and the risk of cardiovascular and all-cause death**. *J Intern Med* 2007, **262**(2):263-272.
- 3. Laukkanen JA, Rauramaa R, Kurl S: Exercise workload, coronary risk evaluation and the risk of cardiovascular and all-cause death in middle-aged men. European journal of cardiovascular prevention and rehabilitation: official journal of the European Society of Cardiology, Working

EudraCT: 2018-002365-19 27<sup>TH</sup> of August 2018

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: \_\_\_\_\_ Journal nr: 2018061692

Groups on Epidemiology & Prevention and Cardiac Rehabilitation and Exercise Physiology 2008, **15**(3):285-292.

- 4. Blair SN, Kohl HW, 3rd, Paffenbarger RS, Jr., Clark DG, Cooper KH, Gibbons LW: **Physical fitness and all-cause mortality. A prospective study of healthy men and women**. *JAMA : the journal of the American Medical Association* 1989, **262**(17):2395-2401.
- 5. Blair SN, Kampert JB, Kohl HW, 3rd, Barlow CE, Macera CA, Paffenbarger RS, Jr., Gibbons LW: Influences of cardiorespiratory fitness and other precursors on cardiovascular disease and all-cause mortality in men and women. *JAMA*: the journal of the American Medical Association 1996, 276(3):205-210.
- 6. Wu T, Gao X, Chen M, van Dam RM: Long-term effectiveness of diet-plus-exercise interventions vs. diet-only interventions for weight loss: a meta-analysis. Obesity reviews: an official journal of the International Association for the Study of Obesity 2009, 10(3):313-323.
- 7. Creel DB, Schuh LM, Reed CA, Gomez AR, Hurst LA, Stote J, Cacucci BM: A randomized trial comparing two interventions to increase physical activity among patients undergoing bariatric surgery. Obesity (Silver Spring) 2016, 24(8):1660-1668.
- 8. Crisp AH, Verlengia R, Ravelli MN, Junior IR, de Oliveira MRM: **Changes in Physical Activities and Body Composition after Roux-Y Gastric Bypass Surgery**. *Obes Surg* 2017.
- 9. King WC, Bond DS: The importance of preoperative and postoperative physical activity counseling in bariatric surgery. *Exercise and sport sciences reviews* 2013, **41**(1):26-35.
- Mundbjerg LH, Stolberg CR, Cecere S, Bladbjerg EM, Funch-Jensen P, Gram B, Juhl CB: Supervised Physical Training Improves Weight Loss After Roux-en-Y Gastric Bypass Surgery: A Randomized Controlled Trial. Obesity (Silver Spring, Md) 2018, 26(5):828-837.
- 11. Stolberg CR, Mundbjerg LH, Funch-Jensen P, Gram B, Bladbjerg EM, Juhl CB: Effects of gastric bypass surgery followed by supervised physical training on inflammation and endothelial function: A randomized controlled trial. *Atherosclerosis* 2018, 273:37-44.
- 12. Stolberg CR, Mundbjerg LH, Funch-Jensen P, Gram B, Juhl CB, Bladbjerg EM: Effects of gastric bypass followed by a randomized study of physical training on markers of coagulation activation, fibrin clot properties, and fibrinolysis. Surg Obes Relat Dis 2018.
- 13. Whitlock EP, Orleans CT, Pender N, Allan J: **Evaluating primary care behavioral counseling interventions: an evidence-based approach**. *Am J Prev Med* 2002, **22**(4):267-284.
- 14. Flegal KM, Kit BK, Orpana H, Graubard BI: **Association of all-cause mortality with overweight and obesity using standard body mass index categories: a systematic review and meta-analysis**. *JAMA : the journal of the American Medical Association* 2013, **309**(1):71-82.
- 15. Lee WJ, Chong K, Chen JC, Ser KH, Lee YC, Tsou JJ, Chen SC: **Predictors of diabetes remission after bariatric surgery in Asia**. *Asian J Surg* 2012, **35**(2):67-73.
- 16. Chaston TB, Dixon JB, O'Brien PE: **Changes in fat-free mass during significant weight loss: a systematic review**. *Int J Obes (Lond)* 2007, **31**(5):743-750.
- 17. Carey DG, Pliego GJ, Raymond RL, Skau KB: **Body composition and metabolic changes following bariatric surgery: effects on fat mass, lean mass and basal metabolic rate**. *Obesity surgery* 2006, **16**(4):469-477.
- 18. Katsanos CS, Madura JA, 2nd, Roust LR: **Essential amino acid ingestion as an efficient nutritional strategy for the preservation of muscle mass following gastric bypass surgery**. *Nutrition (Burbank, Los Angeles County, Calif)* 2016, **32**(1):9-13.
- 19. Yu EW, Bouxsein ML, Putman MS, Monis EL, Roy AE, Pratt JS, Butsch WS, Finkelstein JS: **Two-year changes in bone density after Roux-en-Y gastric bypass surgery**. *The Journal of clinical endocrinology and metabolism* 2015, **100**(4):1452-1459.
- 20. Fleischer J, Stein EM, Bessler M, Della Badia M, Restuccia N, Olivero-Rivera L, McMahon DJ, Silverberg SJ: **The decline in hip bone density after gastric bypass surgery is associated with**

EudraCT: 2018-002365-19 27<sup>TH</sup> of August 2018

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074
Godkendt LMS: Journal nr: 2018061692

**extent of weight loss**. The Journal of clinical endocrinology and metabolism 2008, **93**(10):3735-3740.

- 21. Shanbhogue VV, Stoving RK, Frederiksen KH, Hanson S, Brixen K, Gram J, Jorgensen NR, Hansen S: Bone structural changes after gastric bypass surgery evaluated by HR-pQCT: a two-year longitudinal study. European journal of endocrinology / European Federation of Endocrine Societies 2017, 176(6):685-693.
- 22. Korner J, Punyanitya M, Taveras C, McMahon DJ, Kim HJ, Inabnet W, Bessler M, Gallagher D: **Sex differences in visceral adipose tissue post-bariatric surgery compared to matched non-surgical controls**. *Int J Body Compos Res* 2008, **6**(3):93-99.
- 23. Strain GW, Ebel F, Honohan J, Gagner M, Dakin GF, Pomp A, Gallagher D: **Fat-free mass is not lower 24 months postbariatric surgery than nonoperated matched controls**. *Surg Obes Relat Dis* 2017, **13**(1):65-69.
- 24. Srinivas-Shankar U, Roberts SA, Connolly MJ, O'Connell MD, Adams JE, Oldham JA, Wu FC: Effects of testosterone on muscle strength, physical function, body composition, and quality of life in intermediate-frail and frail elderly men: a randomized, double-blind, placebo-controlled study. The Journal of clinical endocrinology and metabolism 2010, 95(2):639-650.
- 25. Isidori AM, Giannetta E, Greco EA, Gianfrilli D, Bonifacio V, Isidori A, Lenzi A, Fabbri A: **Effects of testosterone on body composition, bone metabolism and serum lipid profile in middle-aged men:** a meta-analysis. *Clinical endocrinology* 2005, **63**(3):280-293.
- 26. Luconi M, Samavat J, Seghieri G, Iannuzzi G, Lucchese M, Rotella C, Forti G, Maggi M, Mannucci E: Determinants of testosterone recovery after bariatric surgery: is it only a matter of reduction of body mass index? Fertility and sterility 2013, 99(7):1872-1879 e1871.
- 27. Pellitero S, Olaizola I, Alastrue A, Martinez E, Granada ML, Balibrea JM, Moreno P, Serra A, Navarro-Diaz M, Romero R *et al*: **Hypogonadotropic hypogonadism in morbidly obese males is reversed after bariatric surgery**. *Obes Surg* 2012, **22**(12):1835-1842.
- 28. Boonchaya-Anant P, Laichuthai N, Suwannasrisuk P, Houngngam N, Udomsawaengsup S, Snabboon T: Changes in Testosterone Levels and Sex Hormone-Binding Globulin Levels in Extremely Obese Men after Bariatric Surgery. *International journal of endocrinology* 2016, **2016**:1416503.
- 29. Ng Tang Fui M, Prendergast LA, Dupuis P, Raval M, Strauss BJ, Zajac JD, Grossmann M: **Effects of testosterone treatment on body fat and lean mass in obese men on a hypocaloric diet: a randomised controlled trial**. *BMC medicine* 2016, **14**(1):153.
- 30. Basaria S, Coviello AD, Travison TG, Storer TW, Farwell WR, Jette AM, Eder R, Tennstedt S, Ulloor J, Zhang A *et al*: **Adverse events associated with testosterone administration**. *The New England journal of medicine* 2010, **363**(2):109-122.
- 31. Whitsel EA, Boyko EJ, Matsumoto AM, Anawalt BD, Siscovick DS: Intramuscular testosterone esters and plasma lipids in hypogonadal men: a meta-analysis. *The American journal of medicine* 2001, 111(4):261-269.
- 32. Fernandez-Balsells MM, Murad MH, Lane M, Lampropulos JF, Albuquerque F, Mullan RJ, Agrwal N, Elamin MB, Gallegos-Orozco JF, Wang AT *et al*: Clinical review 1: Adverse effects of testosterone therapy in adult men: a systematic review and meta-analysis. *The Journal of clinical endocrinology and metabolism* 2010, **95**(6):2560-2575.
- 33. Haider A, Yassin A, Doros G, Saad F: Effects of long-term testosterone therapy on patients with "diabesity": results of observational studies of pooled analyses in obese hypogonadal men with type 2 diabetes. *International journal of endocrinology* 2014, 2014:683515.
- 34. Xu Y, Sun Z: Molecular basis of Klotho: from gene to function in aging. *Endocr Rev* 2015, **36**(2):174-193.

EudraCT: 2018-002365-19 27<sup>TH</sup> of August 2018

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: \_\_\_\_\_ Journal nr: 2018061692

35. Semba RD, Cappola AR, Sun K, Bandinelli S, Dalal M, Crasto C, Guralnik JM, Ferrucci L: **Plasma klotho and mortality risk in older community-dwelling adults**. *The journals of gerontology Series A, Biological sciences and medical sciences* 2011, **66**(7):794-800.

- 36. Glintborg D, Sidelmann JJ, Altinok ML, Mumm H, Andersen M: Increased thrombin generation in women with polycystic ovary syndrome: A pilot study on the effect of metformin and oral contraceptives. *Metabolism: clinical and experimental* 2015, **64**(10):1272-1278.
- 37. Agledahl I, Brodin E, Svartberg J, Hansen JB: Impact of long-term testosterone treatment on plasma levels of free TFPI and TF-induced thrombin generation ex vivo in elderly men with low testosterone levels. *Thromb Haemost* 2009, **102**(5):945-950.
- 38. Glueck CJ, Wang P: **Testosterone therapy, thrombosis, thrombophilia, cardiovascular events**. *Metabolism: clinical and experimental* 2014, **63**(8):989-994.
- 39. Brodin E, Vikan T, Hansen JB, Svartberg J: **Testosterone**, **hemostasis**, **and cardiovascular diseases in men**. *Semin Thromb Hemost* 2011, **37**(1):87-94.
- 40. Bujalska IJ, Kumar S, Stewart PM: **Does central obesity reflect "Cushing's disease of the omentum"?** *Lancet* 1997, **349**(9060):1210-1213.
- 41. Nielsen TL, Hagen C, Wraae K, Brixen K, Petersen PH, Haug E, Larsen R, Andersen M: Visceral and subcutaneous adipose tissue assessed by magnetic resonance imaging in relation to circulating androgens, sex hormone-binding globulin, and luteinizing hormone in young men. The Journal of clinical endocrinology and metabolism 2007, 92(7):2696-2705.
- 42. Sundhedsstyrelsen: National Klinisk Retningslinje for Fedmekirurgi. 2017.
- 43. Mechanick JI, Youdim A, Jones DB, Garvey WT, Hurley DL, McMahon MM, Heinberg LJ, Kushner R, Adams TD, Shikora S *et al*: Clinical practice guidelines for the perioperative nutritional, metabolic, and nonsurgical support of the bariatric surgery patient--2013 update: cosponsored by American Association of Clinical Endocrinologists, the Obesity Society, and American Society for Metabolic & Bariatric Surgery. *Endocrine practice: official journal of the American College of Endocrinology and the American Association of Clinical Endocrinologists* 2013, 19(2):337-372.
- 44. Essendrop M SB, Hansen K: **Reliability of isometric muscle strength tests for the trunk, hands and shoulders**. *Int J Ind Ergonomics* 2001, **28(6)**:379-387.
- 45. Astrand PO RI: A nomogram for calculation of aerobic capacity (physical fitness) from pulse rate during submaximal work. *J Appl Physiol* 1954, **7**(2):218–221.
- 46. Kvorning T, Christensen LL, Madsen K, Nielsen JL, Gejl KD, Brixen K, Andersen M: **Mechanical** muscle function and lean body mass during supervised strength training and testosterone therapy in aging men with low-normal testosterone levels. *Journal of the American Geriatrics Society* 2013, **61**(6):957-962.

### **APPENDIX**

### Adverse reactions/side effects, testosterone.

| System Organ Class | Common | Uncommon | Rare |
|---|---|---|---|
| System Organ Class | $(\geq 1/100 \text{ to} < 1/10)$ | $(\geq 1/1,000 \text{ to } \leq 1/100)$ | $(\geq 1/10,000 \text{ to} <$ |
| | | | 1/1,000) |

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: \_\_\_\_\_ Journal nr: 2018061692

| Blood and lymphatic system disorders | Polycythaemia Haematocrit increased Red blood cell count increased Haemoglobin increased | |
|---|---|---|
| Immune system disorders | | Hypersensibility |
| Metabolism and nutrition disorders | Weight increased | Increased appetite Glycosylated haemoglobin increased Hypercholesterolaemia Blood triglycerides increased Blood cholesterol increased |
| Psychiatric disorders | | Depression Emotional disorder Insomnia Restlessness Aggression Irritability |
| Nervous system disorders | | Headache<br>Migraine<br>Tremor |
| Vascular disorders | Hot flush | Cardiovascular disorder Hypertension Dizziness |
| Respiratory, thoracic and mediastinal disorders | | Bronchitis Sinusitis Cough Dyspnoea |

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: \_\_\_\_\_ Journal nr: 2018061692

| | | Snoring Dysphonia |
|---|---|---|
| Gastrointestinal | | Diarrhoea |
| disorders | | Nausea |
| | | Liver function test |
| | | abnormal |
| Hepatobiliary disorders | | Aspartate |
| | | aminotransferase |
| | | increased |
| | | Alopecia |
| Skin and subcutaneous | | Erythema |
| tissue disorders | Acne | Rash |
| tissue disorders | | Pruritus |
| | | Dry skin |
| | | Arthralgia |
| | | Myalgia |
| Musculoskeletal and | | Pain in extremity |
| connective tissue | | Musculoskeletal |
| disorders | | stiffness |
| disorders | | Blood creatine |
| | | phosphokinase |
| | | increased |
| | | Urine flow decreased |
| Renal and urinary | | Urinary retention |
| disorders | | Urinary tract disorder |
| districts | | Nocturia |
| | | Dysuria |
| Reproductive system | Prostate specific antigen Prostatic intraepithelial | |
| and breast disorders | increased | neoplasia |

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: \_\_\_\_\_ Journal nr: 2018061692

| | Prostate examination | Prostate induration | |
|---|---|---|---|
| | abnormal | Prostatitis | |
| | Benign prostate | Prostatic disorder | |
| | hyperplasia | Libido changes | |
| | | Testicular pain | |
| | | Breast induration | |
| | | Breast pain | |
| | | Gynaecomastia | |
| | | Oestradiol increased | |
| | | Testosterone increased | |
| Canaral digardars and | Various kinds of | Fatigue | |
| General disorders and | Various kinds of | Asthenia | |
| administration site | injection site reactions <sup>1</sup> | Hyperhidrosis | |
| conditions | | Night sweats | |
| Injury, poisoning and | | | Dulmonary oil |
| procedural | | | Pulmonary oil microembolism <sup>2</sup> |
| complications | | | microemoonsm |

<sup>&</sup>lt;sup>1</sup> - Various kinds of injection site reaction: Injection site pain, Injection site discomfort, Injection site pruritus, Injection site erythema, Injection site haematoma, Injection site irritation, Injection site reaction

Other: nervousness, hostility, sleep apnoea, various skin reactions including seborrhea, increased hair growth, increased frequency of erections and in very rare cases jaundice have been reported under treatment with testosterone containing preparations.

Therapy with high doses of testosterone preparations commonly reversibly interrupts or reduces spermatogenesis, thereby reducing the size of the testicles; testosterone replacement therapy of hypogonadism can in rare cases cause persistent, painful erections (priapism). High-dosed or long-

<sup>&</sup>lt;sup>2</sup> - can in rare cases lead to signs and symptoms such as cough, dyspnoea, malaise, hyperhidrosis, chest pain, dizziness, paraesthesia, or syncope. These reactions may occur during or immediately after the injections and are reversible.

EudraCT: 2018-002365-19 27<sup>TH</sup> of August 2018

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074 Godkendt LMS: \_\_\_\_\_ Journal nr: 2018061692

term administration of testosterone occasionally increases the occurrences of water retention and edema.

See SPC for complete safety reference information

(https://www.medicines.org.uk/emc/product/3873/smpc)

EudraCT: 2018-002365-19

Godkendt VEK: \_\_\_\_\_ Projekt ID: S-20180074

Godkendt LMS: Journal nr: 2018061692

## **Counselling intervention**

The overall aim with the counselling is to prevent significant decrease in muscle strength as a consequence of Bariatric surgery. The partial aims are, through counselling, to make the patients aware of the importance of maintaining physical function to increase motivation and PA levels. The Counselling:

The patients will be offered counselling four times during the study period; one exercise counselling before the surgery and three times exercise counselling post-surgery (Table 1). The structure of the counselling will be based on the five A's (Assess, Advise, Agree, Assist, Arrange) however, specific emphasis will be on motivational interviewing, goal setting, individual tailored PA programs, and instructions in the provided programs.

| | Test manual - The effect of testosterone on bodyweight and muscle<br>strength in obese, hypogonadal men undergoing bariatric surgery |
|---|---|
| | Ankomst: |
| | Har forsøgspersonen underskrevet samtykkeerklæring? Kort introduktion om hvad der skal foregå. Montering af accelerometer |
| PDF with test protocol (double-click to open) | Cand Scient I Idraet og Sundhed, Ph.d. Båld Gram |